CLINICAL TRIAL: NCT01877538
Title: "[11C]Donepezil PET for Imaging the Parasympathetic Nervous System in Healthy Adults"
Brief Title: Study to Investigate the Ability of [11C]Donepezil PET to Image the Parasympathetic Nervous System
Status: Completed | Type: Observational
Sponsor: Per Borghammer (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Sponsor-Investigator, Per Borghammer, MD, PhD, DMSci, Aarhus University Hospital
Organization: University of Aarhus (Other)
Other Study IDs: 01-01
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- [11C]donepezil PET: [11C]donepezil is a radiopharmaceutical. It is evaluated whether the binding of [11C]donepezil in various peripheral tissues is in accordance with known distribution of the parasympathetic nervous system.
  Interventions: Other: [11C]donepezil PET

INTERVENTIONS:
Other: [11C]donepezil PET — Positron Emission Tomography (PET) imaging of acetylcholinesterase with the ligand [11C]donepezil

SUMMARY:
AIM: To validate the tracer [11C]donepezil for use in the parasympathetic nervous system.

MATERIALS AND METHODS: The Investigators will include 7 healthy males aged 45-75 in our study. The participants will receive a careful medical examination, including a neurological examination, as part of the inclusion process. The subjects also have an MRI scan of the brain. PET/CT scans with [11C]donepezil are conducted. Six subjects will receive two PET/CT scans - once for the upper abdominal region and once for the head region two evaluate dynamic binding characteristics of the tracer in internal organ. Additionally, one single subject will receive 5 consecutive whole body PET scans to estimate radioactive dosimetry of this tracer.

PERSPECTIVES: The study will potentially result in the development of a PET ligand for imaging the parasympathetic nervous system. This will have applications for research in Parkinson's disease, diabetes, heart disease and other disorders, in which the autonomic nervous system is involved

DETAILED DESCRIPTION:
Please see the published paper wherein all details are listed:

In vivo imaging of human acetylcholinesterase density in peripheral organs using 11C-donepezil: dosimetry, biodistribution, and kinetic analyses.

Gjerløff T, Jakobsen S, Nahimi A, Munk OL, Bender D, Alstrup AK, Vase KH, Hansen SB, Brooks DJ, Borghammer P. J Nucl Med. 2014 Nov;55(11):1818-24.

ELIGIBILITY:
Inclusion Criteria:

* male
* 45-75 years

Exclusion Criteria:

* dementia,
* psychiatric diseases,
* serious medical illness including any type of previous cancer, any drug with known interaction with the autonomic nervous system

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 7 healthy male volunteers is included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Borghammer, MD,PhD, Principal Investigator — Dept. of Nuclear Medicine & PET Center, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Dep. of Nuclear Medicine and PET centre, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gjerloff T, Jakobsen S, Nahimi A, Munk OL, Bender D, Alstrup AK, Vase KH, Hansen SB, Brooks DJ, Borghammer P. In vivo imaging of human acetylcholinesterase density in peripheral organs using 11C-donepezil: dosimetry, biodistribution, and kinetic analyses. J Nucl Med. 2014 Nov;55(11):1818-24. doi: 10.2967/jnumed.114.143859. Epub 2014 Oct 16. PMID 25324520

RESULTS

PARTICIPANT FLOW:
Groups:
- [11C]Donepezil: [11C]donepezil is a radiopharmaceutical. It is evaluated whether the binding in peripheral tissues is in accordance with known distribution of the parasympathetic nervous system
  [11C]donepezil PET: Positron Emission Tomography (PET) imaging of acetylcholinesterase with the ligand [11C]donepezil
  7 healthy control subjects were scanned in this preliminary pilot study.
Period: Overall Study
Arm/Group | [11C]Donepezil
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 7 healthy control subjects
Groups:
- [11C]Donepezil PET: [11C]donepezil is a radiopharmaceutical used with Positron Emission Tomography (PET) imaging. It is evaluated whether the binding in peripheral tissues is in accordance with known distribution of the parasympathetic nervous system
  [11C]donepezil PET: Positron Emission Tomography (PET) imaging of acetylcholinesterase with the ligand [11C]donepezil
  7 healthy control subjects were recruited to this study.
Arm/Group | [11C]Donepezil PET
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Distribution Volume (DV) of [11C]Donepezil - BASELINE
Description: Logan's graphical analysis is used to calculate Distribution Volumes in Volumes of interest in internal organs (salivary gland, heart, liver, stomach, intestines, kidneys). Arterial blood sampling with radio metabolite correction is performed.
Time Frame: 1 day (One timepoint)
Population: In 6 subjects we analysed Volumes of distribution (Vd) and SUV values in internal organs (parotid, submandibular, spleen, stomach, heart, intestine, pancreas). NOTE: In subject number 7 we examined radioactive dose in 23 target organs (dose: microSv/MBq) and calculated the combined effective dose. The Vd and SUV values listed are from 6 subjects.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- [11C]Donepezil PET: [11C]donepezil is a radiopharmaceutical. It is evaluated whether the binding in peripheral tissues is in accordance with known distribution of the parasympathetic nervous system
  [11C]donepezil PET: Positron Emission Tomography (PET) imaging of acetylcholinesterase with the ligand [11C]donepezil
Arm/Group | [11C]Donepezil PET
Number analyzed (Participants) | 6
mL
  Vd - Parotid | 18.0 (3.3)
  Vd - Submandibular | 22.1 (5.0)
  Vd - Spleen | 21.4 (7.6)
  Vd - Stomach | 26.6 (11.5)
  Vd - Heart | 46.8 (7.8)
  Vd - Intestine | 103.9 (19.5)
  Vd - Pancreas | 189.8 (103.9)

2. Primary Outcome: Standard Uptake Value (SUV) of [11C]Donepezil - BASELINE
Description: SUV values were calculated in 7 internal organs. SUV is a unitless ratio. We normalised to injected dose and bodyweight.
  SUV (organ) = activity concentration (organ; kBq/mL) * bodyweight (mL) / injected dose (kBq)
  Note: it is a common assumption when calculating SUV values that bodyweight equals volume, and therefore the unit mL is appropriate.
Time Frame: 1 day (one timepoint)
Population: In 6 subjects the SUV values in internal organs were calculated.
Measure: Mean (Standard Deviation); unit: Unitless ratio
Arm/Group | [11C]Donepezil PET
Number analyzed (Participants) | 6
Unitless ratio
  SUV - Parotid | 2.3 (0.5)
  SUV - Submandibular | 3.9 (1.1)
  SUV - Spleen | 3.7 (1.4)
  SUV - Stomach | 4.8 (1.2)
  SUV - Heart | 7.4 (0.8)
  SUV - Intestine | 11.7 (2.4)
  SUV - Pancreas | 19.1 (4.2)

ADVERSE EVENTS:
Groups:
- [11C]Donepezil: [11C]donepezil is a radiopharmaceutical. It is evaluated whether the binding in peripheral tissues is in accordance with known distribution of the parasympathetic nervous system
  [11C]donepezil PET: Positron Emission Tomography (PET) imaging of acetylcholinesterase with the ligand [11C]donepezil
  7 healthy controls were PET scanned in this preliminary study.
  No adverse events were detected.
Arm/Group | [11C]Donepezil
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No